CLINICAL TRIAL: NCT06650475
Title: Evaluation of the Optic Nerve Sheath Diameter in Children Undergoing Laparoscopic Abdominal Surgery at Low and Standard Gas Insufflation Pressures
Brief Title: "Optic Nerve Sheath Diameter; Low vs. Conventional Insufflation Pressures''
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Yasin Tire, MD, Anesthesiologist, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Study Pedlap
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: ONSD in Laparoscopic Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low pressure (Active Comparator): Group L will undergo laparoscopy under low pressure (8-10mm Hg).
  Interventions: Procedure: Using low or standart pressure
- Standart Pressure (Sham Comparator): Standard pressures (12-16 mmHg) are used in laparoscopic surgery for patients in Group S.
  Interventions: Procedure: Using low or standart pressure

INTERVENTIONS:
Procedure: Using low or standart pressure — Written consent will be obtained before the randomized study. Randomization will be done on the computer using a software program. Participants will be divided into two groups. Patients in Group S will undergo laparoscopy under standard pressures (12-16 mmHg) in laparoscopic surgery, while patients in Group L will undergo laparoscopy under low pressure (8-10 mm Hg).

SUMMARY:
Objective: This study investigates the impact of carbon dioxide (CO2) pneumoperitoneum on optic nerve sheath diameter (ONSD) and intracranial pressure (ICP) in patients undergoing total laparoscopic hysterectomy. Previous research suggests that pneumoperitoneum can lead to elevated ICP, with the standard intracranial monitoring technique being invasive intraventricular catheter placement. In contrast, bedside ultrasound assessment of ONSD offers a noninvasive alternative for detecting increased ICP.

Methods: The Hypothesize will be standard gas insufflation pressure significantly increases ONSD, while low-pressure insufflation will maintain ONSD levels. The primary aim is to compare ONSD variations pre- and post-CO2 insufflation in patients subjected to both low-pressure and standard-pressure laparoscopic surgery. Secondary aims include evaluating end-tidal CO2 measurements between the two groups.

DETAILED DESCRIPTION:
It has been shown in many studies that pneumoperitoneum containing carbon dioxide (CO2) during laparoscopy increases intracranial pressure (ICP). (1) Evaluation of the Effect of Intraabdominal Pressure on Optic Nerve Sheath Diameter in Patients Undergoing Total Laparoscopic Hysterectomy. The standard technique for monitoring ICP is the placement of an intraventricular catheter connected to an external pressure transducer. (2) Bedside evaluation of optic nerve sheath diameter (ONSD) with ultrasound technique is a more practical and noninvasive method used to determine high ICP (>20 mmHg). The anatomical continuity of the dura with the optic nerve sheath (ONSD) allows the use of this technology, and thus an increase in ICP can be transmitted from the subarachnoid space to the ONSD. (3)

Low-pressure pneumoperitoneum reduces analgesic consumption after laparoscopic cholecystectomy in studies, but the effect of standard and low intraabdominal pressures on ICP has not yet been clarified. (4)

In our thesis, assuming that standard gas insufflation pressure will increase ONSD, but low gas insufflation pressure will not cause a change, the primary aim was to compare ONSD between two groups of low-pressure and standard-pressure laparoscopic surgery before and after CO2 insufflation preoperatively. Second, the end-tidal CO2 measurements between the two groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted in patients under 18 years of age with American Society of Anesthesiologists (ASA) I-II.

Exclusion Criteria:

* Patients with a history of neurological disease, glaucoma, surgery exceeding 2 hours, known chronic obstructive pulmonary disease (COPD), heart disease, and previous lung surgery will be excluded from the study. Patients with intraoperative hemodynamic problems; ETCO2 greater than 45 mmHg, plateau pressure over 30 cmH2, and peak inspiratory pressure over 35 cmH2 will be excluded from the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | 5 min after intubation (T1). Intra-abdominal 10 min (T2) and 10 min after positioning (T3)
  For the measurement of ONSD (Optic Nerve Sheath Diameter) a portable, software controlled, ultrasonographic system (Micromax Ultrasound System, SonoSitelnc. Bothell, Washington, USA) 13-6 MHz 38 mm wide band linear array transducer will be used. The probe positioning will be done in the axial plane over the closed eye and ONSD will be determined by the two hyperechoic lines on the back. The outer limits will be determined by electronic calipers as hyperechoic lines behind the 3 papillae. Measurements will be taken from each eye in all patients. In order to neutralize the intraoperative variability, the average of these measurements will be taken.

SECONDARY OUTCOMES:
CO2 measurements | after 5 minutes (T1) 10 minutes (T2), 10 minutes after position (T3)
  Secondary will be the evaluation of end tidal CO2 measurements between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Tire, Assoc. Prof., Study Director — Konya City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Konya City Hospital, Konya, Meram
  - Yasin Tire, Konya, Meram